CLINICAL TRIAL: NCT05299905
Title: Developing Immersive Gamification Technology System (ImGTS) for Rehabilitation Management of Pediatric Patients With Cerebral Palsy and With Mobility Limitations (Phase 1 Trial)
Brief Title: ImGTS for Patients With Cerebral Palsy and With Mobility Limitations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augmented eXperience E-health Laboratory (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AXEL0002
Record Dates: First submitted 2022-02-06; First posted 2022-03-29 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2022-03

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semi-CAVE (Experimental)
  Interventions: Procedure: Virtual reality using Semi-CAVE
- Head-mounted display system (Experimental)
  Interventions: Procedure: Virtual reality using the HMD

INTERVENTIONS:
Procedure: Virtual reality using Semi-CAVE — The Semi-CAVE will use two screens positioned at a corner of the room, each with a ceiling-mounted short throw projector in front. The participant will stand in the middle of the area, giving them a viewing angle of roughly 180 degrees. The participant will be wearing a safety harness secured to an overhead guide rail, if necessary. The participant may be standing freely, on a treadmill, or on a step stool depending on the type of activity to be performed. The participant will interact with the system through motion sensors positioned at the corners of the area. To one side of the area will be a sufficiently powerful computer running the software. The projectors will be connected to this computer via HDMI cables or similar.
  Arms: Semi-CAVE
Procedure: Virtual reality using the HMD — The HMD will be a commercially available device that uses handheld controllers to control movement while in the VE. The researchers will use a room-scale set-up where a 3 m x 3 m square space is required. Oculus Quest 2 Controllers will be used to interact with the VE. The user will be positioned at the center of the square by default. A therapist will assist them through a separate program called the Observation Module. This program will let the therapist view what the patient can see in the HMD. This will also be used by the therapist to guide the patient navigate through the VE and give instructions for the activities.
  Arms: Head-mounted display system

SUMMARY:
The proposed research project aims to answer the question "Are immersive technology systems effective in the rehabilitation management of pediatric patients with cerebral palsy and with mobility limitations?". The current study is the first of three phases, and it aims to create an immersive gamification technology system for the management of patients with cerebral palsy and with mobility disorders and to determine its acceptability, usability, and safety in healthy children.

DETAILED DESCRIPTION:
The participants will undergo an intervention using the assigned ImGTS for four sessions (twice a week for two weeks) for at most 1 hour per session. The experience will last for at most 20 minutes, interspersed with 5- to 20-minute breaks. The researchers will document the participants' reaction and interaction with the ImGTS. Participants will be staying at the designated laboratory for not more than one hour.

Demographic characteristics of the participant (age, sex, educational level, primary caregiver, list of medications, hobbies and interests, previous experience with VR applications, existing illnesses and medications) will be collected through an interview with the child and the participant's parent, legal guardian, or caregiver.

Safety will be determined by assessing a participant's experience of cybersickness using a cybersickness questionnaire that will be administered before and after each session. In this self-report questionnaire, nine symptoms will be rated as absent/none, slight, moderate, or severe. These symptoms are general discomfort, fatigue, eyestrain, difficulty focusing, headache, fullness of head, blurred vision, dizziness when the eyes are closed, and vertigo. The questionnaire will take around 10 minutes to complete. If a participant will experience severe cybersickness, the participant may opt to discontinue the experience. The participant will be instructed to remove the HMD or to step out of the Semi-CAVE room to rest and recover from the symptoms. A medical professional will be present to monitor the participant's symptoms and to attend to the participant for further management. The reason(s) for discontinuing the experience will be documented.

The acceptability of the design will be measured using the Place Probe, a sense of place questionnaire. The questionnaire will be administered after each session, and it will collect information on a participant's experience in the VR application, particularly on (1) general impression of the environment, (2) the key features of the environment, and (3) feelings of presence. A positive general impression, a memorable environment, and a high level of presence will indicate that the VE developed is acceptable. This will take about 10 minutes to complete.

Usability testing will be performed according to the PNS ISO/IEC Metrics. The goal is to provide continuous improvement in the design and user experience to maximize the three components of usability: effectiveness, efficiency, and satisfaction. Additional usability metrics will be identified during the first phase of the study. The metrics will be specifically adjusted to the target participants as well as the contents to be included in the ImGTS.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 to 12 years old
* Demonstrates fine and gross motor abilities within the norm for the child's age as measured by the Bruininks-Oseretsky Test of Motor Proficiency Test (BOTMP)

Exclusion Criteria:

* Previously diagnosed with any developmental disorder including CP
* Has had episodes of seizures or previously diagnosed as having epilepsy
* Has a history of motion sickness
* Unable to follow one-step instructions

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Number of participants with 'Moderate' or 'Severe' symptoms of cybersickness as assessed by the Virtual Reality Sickness Questionnaire before Session 1 | Immediately before Session 1, within an hour of before use of the virtual reality game
  Baseline assessment for the presence of cybersickness symptoms for Session 1 will be done using the Virtual Reality Sickness Questionnaire. The questionnaire uses a 4-point scale (None, Slight, Moderate, Severe) to assess nine symptoms of cybersickness. More 'Severe' symptoms mean lower safety.
Number of participants with 'Moderate' or 'Severe' symptoms of cybersickness as assessed by the Virtual Reality Sickness Questionnaire after Session 1 | Immediately after Session 1, within an hour of completion of the virtual reality game
  Assessment for the occurrence of cybersickness symptoms for Session 1 will be done using the Virtual Reality Sickness Questionnaire. The questionnaire uses a 4-point scale (None, Slight, Moderate, Severe) to assess nine symptoms of cybersickness. More 'Severe' symptoms mean lower safety.
Number of participants with 'Moderate' or 'Severe' symptoms of cybersickness as assessed by the Virtual Reality Sickness Questionnaire before Session 2 | Immediately before Session 2, within an hour of before use of the virtual reality game
  Baseline assessment for the presence of cybersickness symptoms for Session 2 will be done using the Virtual Reality Sickness Questionnaire. The questionnaire uses a 4-point scale (None, Slight, Moderate, Severe) to assess nine symptoms of cybersickness. More 'Severe' symptoms mean lower safety.
Number of participants with 'Moderate' or 'Severe' symptoms of cybersickness as assessed by the Virtual Reality Sickness Questionnaire after Session 2 | Immediately after Session 2, within an hour of completion of the virtual reality game
  Assessment for the occurrence of cybersickness symptoms for Session 2 will be done using the Virtual Reality Sickness Questionnaire. The questionnaire uses a 4-point scale (None, Slight, Moderate, Severe) to assess nine symptoms of cybersickness. More 'Severe' symptoms mean lower safety.
Number of participants with 'Moderate' or 'Severe' symptoms of cybersickness as assessed by the Virtual Reality Sickness Questionnaire before Session 3 | Immediately before Session 3, within an hour of before use of the virtual reality game
  Baseline assessment for the presence of cybersickness symptoms for Session 3 will be done using the Virtual Reality Sickness Questionnaire. The questionnaire uses a 4-point scale (None, Slight, Moderate, Severe) to assess nine symptoms of cybersickness. More 'Severe' symptoms mean lower safety.
Number of participants with 'Moderate' or 'Severe' symptoms of cybersickness as assessed by the Virtual Reality Sickness Questionnaire after Session 3 | Immediately after Session 3, within an hour of completion of the virtual reality game
  Assessment for the occurrence of cybersickness symptoms for Session 3 will be done using the Virtual Reality Sickness Questionnaire. The questionnaire uses a 4-point scale (None, Slight, Moderate, Severe) to assess nine symptoms of cybersickness. More 'Severe' symptoms mean lower safety.
Number of participants with 'Moderate' or 'Severe' symptoms of cybersickness as assessed by the Virtual Reality Sickness Questionnaire before Session 4 | Immediately before Session 4, within an hour of before use of the virtual reality game
  Baseline assessment for the presence of cybersickness symptoms for Session 4 will be done using the Virtual Reality Sickness Questionnaire. The questionnaire uses a 4-point scale (None, Slight, Moderate, Severe) to assess nine symptoms of cybersickness. More 'Severe' symptoms mean lower safety.
Number of participants with 'Moderate' or 'Severe' symptoms of cybersickness as assessed by the Virtual Reality Sickness Questionnaire after Session 4 | Immediately after Session 4, within an hour of completion of the virtual reality game
  Assessment for the occurrence of cybersickness symptoms for Session 4 will be done using the Virtual Reality Sickness Questionnaire. The questionnaire uses a 4-point scale (None, Slight, Moderate, Severe) to assess nine symptoms of cybersickness. More 'Severe' symptoms mean lower safety.
The acceptability of the design for Session 1 will be measured using the Place Probe | Immediately after Session 1, within an hour of completion of the virtual reality game
  The Place Probe is a questionnaire that is composed of three parts and measures a person's general impression of a place (qualitative), their perception on key features of a place (quantitative), and their feelings of presence (quantitative), respectively. Under key features of place, the virtual environment will be assessed according to 33 pairs of semantic differentials where more positive answers mean a better outcome. Under feelings of presence, higher mean scores mean higher levels of immersion
The acceptability of the design for Session 2 will be measured using the Place Probe | Immediately after Session 2, within an hour of completion of the virtual reality game
  The Place Probe is a questionnaire that is composed of three parts and measures a person's general impression of a place (qualitative), their perception on key features of a place (quantitative), and their feelings of presence (quantitative), respectively. Under key features of place, the virtual environment will be assessed according to 33 pairs of semantic differentials where more positive answers mean a better outcome. Under feelings of presence, higher mean scores mean higher levels of immersion
The acceptability of the design for Session 3 will be measured using the Place Probe | Immediately after Session 3, within an hour of completion of the virtual reality game
  The Place Probe is a questionnaire that is composed of three parts and measures a person's general impression of a place (qualitative), their perception on key features of a place (quantitative), and their feelings of presence (quantitative), respectively. Under key features of place, the virtual environment will be assessed according to 33 pairs of semantic differentials where more positive answers mean a better outcome. Under feelings of presence, higher mean scores mean higher levels of immersion
The acceptability of the design for Session 4 will be measured using the Place Probe | Immediately after Session 4, within an hour of completion of the virtual reality game
  The Place Probe is a questionnaire that is composed of three parts and measures a person's general impression of a place (qualitative), their perception on key features of a place (quantitative), and their feelings of presence (quantitative), respectively. Under key features of place, the virtual environment will be assessed according to 33 pairs of semantic differentials where more positive answers mean a better outcome. Under feelings of presence, higher mean scores mean higher levels of immersion
Observation of completion of the game in the given time during Session 4 to measure effectiveness of the application | For one hour during Session 4
  Effectiveness is a component of usability, and will be assessed through observing completion of the game within the allotted time. If at least 85% of the participants complete the game within the allotted time, the game is said to be effective.
Observation of ease of use of controls and user interaction during Session 4 to measure efficiency of the application during Session 4 | For one hour during Session 4
  Efficiency is a component of usability that will assess a participant's ease of use of the controls and user interface during the experience. If at least 85% of the participants do not encounter or express difficulties in using the application during the experience, the game is said to be efficient.
Observation of user reactions to measure satisfaction in using the application through during Session 4 | For one hour during Session 4
  Satisfaction is a component of usability that will assess a participant's enjoyment in using the game. It will be assessed through observing the reaction of the participant during Session 4. If 90% of the participants visibly show or verbally express enjoyment during the experience, the game is said to be satisfactory.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Eliza R Aguila, PhD, Principal Investigator — University of the Philippines Manila
Locations (1):
- College of Allied Medical Professions Clinic for Therapy Services, Manila, National Capital Region, Philippines

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Billingham SA, Whitehead AL, Julious SA. An audit of sample sizes for pilot and feasibility trials being undertaken in the United Kingdom registered in the United Kingdom Clinical Research Network database. BMC Med Res Methodol. 2013 Aug 20;13:104. doi: 10.1186/1471-2288-13-104. PMID 23961782
- [Background] Birckhead B, Khalil C, Liu X, Conovitz S, Rizzo A, Danovitch I, Bullock K, Spiegel B. Recommendations for Methodology of Virtual Reality Clinical Trials in Health Care by an International Working Group: Iterative Study. JMIR Ment Health. 2019 Jan 31;6(1):e11973. doi: 10.2196/11973. PMID 30702436
- [Background] Chen Y, Fanchiang HD, Howard A. Effectiveness of Virtual Reality in Children With Cerebral Palsy: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Phys Ther. 2018 Jan 1;98(1):63-77. doi: 10.1093/ptj/pzx107. PMID 29088476
- [Background] Demers M, Fung K, Subramanian SK, Lemay M, Robert MT. Integration of Motor Learning Principles Into Virtual Reality Interventions for Individuals With Cerebral Palsy: Systematic Review. JMIR Serious Games. 2021 Apr 7;9(2):e23822. doi: 10.2196/23822. PMID 33825690
- [Background] Kim HK, Park J, Choi Y, Choe M. Virtual reality sickness questionnaire (VRSQ): Motion sickness measurement index in a virtual reality environment. Appl Ergon. 2018 May;69:66-73. doi: 10.1016/j.apergo.2017.12.016. Epub 2018 Jan 16. PMID 29477332
- [Background] Novak I, McIntyre S, Morgan C, Campbell L, Dark L, Morton N, Stumbles E, Wilson SA, Goldsmith S. A systematic review of interventions for children with cerebral palsy: state of the evidence. Dev Med Child Neurol. 2013 Oct;55(10):885-910. doi: 10.1111/dmcn.12246. Epub 2013 Aug 21. PMID 23962350
- [Background] Paulson A, Vargus-Adams J. Overview of Four Functional Classification Systems Commonly Used in Cerebral Palsy. Children (Basel). 2017 Apr 24;4(4):30. doi: 10.3390/children4040030. PMID 28441773
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Sandlund M, McDonough S, Hager-Ross C. Interactive computer play in rehabilitation of children with sensorimotor disorders: a systematic review. Dev Med Child Neurol. 2009 Mar;51(3):173-9. doi: 10.1111/j.1469-8749.2008.03184.x. Epub 2009 Jan 26. PMID 19191834
- [Background] Smits-Engelsman BC, Blank R, van der Kaay AC, Mosterd-van der Meijs R, Vlugt-van den Brand E, Polatajko HJ, Wilson PH. Efficacy of interventions to improve motor performance in children with developmental coordination disorder: a combined systematic review and meta-analysis. Dev Med Child Neurol. 2013 Mar;55(3):229-37. doi: 10.1111/dmcn.12008. Epub 2012 Oct 29. PMID 23106530
- [Background] Weber H, Barr C, Gough C, van den Berg M. How Commercially Available Virtual Reality-Based Interventions Are Delivered and Reported in Gait, Posture, and Balance Rehabilitation: A Systematic Review. Phys Ther. 2020 Sep 28;100(10):1805-1815. doi: 10.1093/ptj/pzaa123. PMID 32691059
- [Background] Weiss PL, Rand D, Katz N, Kizony R. Video capture virtual reality as a flexible and effective rehabilitation tool. J Neuroeng Rehabil. 2004 Dec 20;1(1):12. doi: 10.1186/1743-0003-1-12. PMID 15679949